CLINICAL TRIAL: NCT06578715
Title: The Effect of Emotional Freedom Technique (EFT) Applied to Postmenopausal Women on Sleep and Quality of Life: A Randomized Controlled Trial
Brief Title: Emotional Freedom Technique (EFT) Applied to Postmenopausal Women on Sleep and Quality of Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aslı SİS ÇELİK, Associate Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: aslı12
Record Dates: First submitted 2024-08-28; First posted 2024-08-29 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Menopause Related Conditions

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): no intervention will be applied to the control group
- Experimental Group (Experimental): EFT will be applied to the women to be included in the experimental group in the study once a week, a total of four times in a month.
  Interventions: Behavioral: Emotional Freedom Technique

INTERVENTIONS:
Behavioral: Emotional Freedom Technique — EFT basically involves serial tapping on acupuncture points, no needles are used, there is no invasive procedure, there are affirmation suggestions, it is an easy, painless, simple but effective method that can be done in minutes. It is realized by applying kinetic energy to certain meridians on the head and chest with the fingertips. The points where the tapping is done are the end points of the meridians in the body. They are located symmetrically on both sides of the body. Since these points are close to the skin surface, they are points that are more easily reached than the deeper buried parts of the meridians. While applying pressure with the fingertips, the individual needs to focus on the problem that bothers him/her. Another thing that needs to be done at the same time is for the person to make positive suggestions to himself/herself vocally.
  Arms: Experimental Group

SUMMARY:
The study will be conducted as a randomized controlled experimental study to determine the effects of the Emotional Freedom Technique (EFT) applied to women in menopause on sleep quality and quality of life.

It will be conducted with 80 women between the ages of 45-64, registered in a family health center in a city in the east of Turkey, who have been in menopause for at least one year and volunteer to participate in the study.

EFT will be applied to the women to be included in the experimental group in the study once a week, a total of four times in a month.

The "Participant Information Form", "Utian Quality of Life Scale" and "Pittsburgh Sleep Quality Scale" prepared by the researchers in line with the literature information will be used in the collection of research data.

DETAILED DESCRIPTION:
The study will be conducted as a randomized controlled experimental study to determine the effects of the Emotional Freedom Technique (EFT) applied to women in menopause on sleep quality and quality of life.

It will be conducted with 80 women between the ages of 45-64, registered in a family health center in a city in the east of Turkey, who have been in menopause for at least one year and volunteered to participate in the study.

The "simple randomization method" will be selected as the randomization method in the study in order to provide an equal number of samples in two groups. A random number table will be created in a computer environment using the httpp://www.randomizer.org/website for the 80 participants to be sampled, with numbers from 1 to 80 in two groups. It will be decided by tossing a coin to determine which group the groups should be in. The names on the list will be evaluated according to the group corresponding to that order in the table, and accordingly, 40 women will be assigned to the experimental group and 40 women will be assigned to the control group.

EFT will be applied to the women to be included in the experimental group in the study once a week, a total of four times in a month.

When the research is completed, the data of the experimental and control groups (coded as X and Y) will be transferred to the computer environment by a statistician independent of the research and the data will be analyzed and the findings will be reported. Our research is planned to be conducted as a single-blind study in which the statistician will be blinded.

The "Participant Information Form", "Utian Quality of Life Scale" and "Pittsburgh Sleep Quality Scale" prepared by the researchers in line with the literature information will be used in the collection of research data.

Pre-Test Data will be collected between September-October 2024, the interim measurement after the EFT intervention will be made between October-November 2024, and the final measurement will be made between November-December 2024.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Being able to read and write in Turkish,
* Women between the ages of 45-64 who have not had menstrual bleeding for at least one year (women under the age of 65 who have entered natural menopause),
* Not being diagnosed with a psychiatric disease,
* Not using Hormone Replacement Therapy (HRT),
* Not using antidepressants, antihistamines, benzodiazepines, hypnotics and narcotics, etc.,
* Not using any complementary and alternative medicine (such as Reiki, phytoestrogens, acupressure).
* Scoring '5 and above' on the Pittsburgh Sleep Quality Scale

Exclusion Criteria:

* Starting to use Hormone Replacement Therapy after starting the study,
* Starting to use antidepressants, antihistamines, benzodiazepines, hypnotics and narcotics, etc.,
* Starting to use any complementary and alternative medicine method,
* Voluntarily leaving the study.

Ages: 45 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life levels during menopause | 1 month
  The difference between the Utian Quality of Life Scale pretest and posttest mean scores of women in both groups. The lowest score that can be obtained from the scale is 23, and the highest score is 115. An increase in the scale score indicates an increase in the quality of life.
Quality of sleep levels during menopause | 1 month
  The difference between the Utian Quality of Life Scale pretest and posttest mean scores of women in both groups. The sleep quality of individuals whose total scale score is 5 points or less is considered "good"; the sleep quality of individuals whose score is above 5 points is considered "bad".

CONTACTS AND LOCATIONS:
Overall Officials: Aslı SİS ÇELİK, Study Director — Ataturk University